CLINICAL TRIAL: NCT01438801
Title: Predictive Value of Baseline and Stimulated Serum IGF-1 and IGFBP-3 During a Dose-escalation IGF-1 Generation Test for the 1 Year Growth Response to Growth Hormone (GH) Therapy in Short Children With Low IGF-1 and a Normal GH Peak in a Provocation Test
Brief Title: Predictive Value of the Insulin-like Growth Factor-1 (IGF-1) Generation Test for the Growth Response to Growth Hormone Treatment (PRED-IGF)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Participant enrollment was not feasible
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A-95-58035-017; 2010-019980-13 (EudraCT Number)
Record Dates: First submitted 2011-08-24; First posted 2011-09-22 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Short Stature
MeSH Terms: interventions — Human Growth Hormone; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NutropinAq (Experimental)
  Interventions: Drug: Nutropin [Somatropin (rDNA origin) for injection]

INTERVENTIONS:
Drug: Nutropin [Somatropin (rDNA origin) for injection] — Doses in the diagnostic protocol are 0.7 and 1.4 mg/m2/day, injected by subcutaneous injection at bedtime for 2 weeks, divided by washout periods of preferably 4 weeks (accepted range 4-6 weeks). An additional period of 2 weeks on 2.8 mg/m2/day (after a washout period of 4-6 weeks) will be added if the IGF-I response on either dosage is insufficient (serum IGF-I SDS <0).

SUMMARY:
The evaluation of a standardized diagnostic test to predict the growth response in a 1 year trial with Growth Hormone (GH) treatment (carried out in the context of regular patient care) in non GH deficient short children with low serum insulin-like growth factor-1 (IGF-1).

ELIGIBILITY:
Inclusion Criteria:

* Age 2.0 - 9.0 years for females, 2.0 - 10.0 yrs for males.
* Prepubertal stage (Tanner 1 for breast (B1) in females, or Tanner 1 for genitals (G1) for males).
* Bone age < 10 'years' (males) or < 9 'years' (females) according to Greulich and Pyle. The bone age will be read by the pediatric endocrinologist responsible for the pre-study screening visit.
* Height SDS < -2.5 for ethnically adequate references. For children of Dutch or Western European origin the 1997 nation-wide references for Dutch children will be used. For children of Moroccan or Turkish origin, the respective reference charts will be used. For children of other ethnicities, the 1977 North American (NCHS/WHO) reference will be used, as these charts have been accepted by WHO as world-wide standard from the age of 5 years.

Exclusion Criteria:

* Has a history of hypersensitivity to growth hormone or phenol (conservative added to GH in NutropinAq), or drugs with a similar chemical structure.
* Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the subject's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.
* Has a birth weight and/or length below -2 SDS for Swedish reference charts. Patients will not be excluded due to an unknown birth weight or length.
* Has a known cause of short stature, or any significant concomitant disease that is likely to interfere with growth or with the study schedule/objectives, or is a known contraindication to GH treatment.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Estimated); Primary Completion 2013-05-31 (Estimated); Study Completion 2013-05-31 (Estimated)

PRIMARY OUTCOMES:
Peak serum IGF-1 level with GH (1.4 mg/m2/day) change from baseline. | Week 2

SECONDARY OUTCOMES:
Delta IGF-1 SDS on 0.7 & 1.4 mg GH/m2/day | Baseline, week 2
Delta insulin-like growth factor binding protein-3 (IGFBP-3) standard deviation score (SDS) on 0.7 & 1.4 mg GH/m2/day | Baseline, week 2
Delta of the ratio IGF-1:IGFBP-3 SDS on 0.7 mg & 1.4 mg GH/m2/day | Baseline, week 2
Delta of the ratio IGF-1:IGFBP-2 (insulin-like growth factor binding protein-2) SDS on 0.7 mg & 1.4 mg GH/m2/day | Baseline, week 2
Peak IGFBP-3 SDS on 0.7 mg & 1.4 mg GH/m2/day | Baseline, week 2
Peak of the ratio IGF-1:IGFBP-3 SDS on 0.7 mg & 1.4 mg GH/m2/day | Baseline, week 2
Peak of the ratio IGF-1:IGFBP-2 SDS on 0.7 mg & 1.4 mg GH/m2/day | Baseline, week 2

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, MD, Study Director — Ipsen